CLINICAL TRIAL: NCT05419154
Title: A Pragmatic, Multi-center, Multi-surgeon Prospective Outcome Study on Immediate Pain-dependent Weight-bearing Without Immobilization After Surgically Treated Ankle Fractures
Brief Title: Full-Weightbearing Following Ankle Fractures Surgically Treated - The FAST-Mobility Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); University Medical Center Rostock (Other); University Hospital Muenster (Other); University Hospital Carl Gustav Carus (Other)
Responsible Party: Principal Investigator, Sebastian. F. Baumbach, Head of Foot and Ankle Department, Assistant Professor, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Weightbearing Ankle Fracture
Record Dates: First submitted 2022-05-30; First posted 2022-06-15 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Rehabilitation of Surgically Treated Ankle Fractures
MeSH Terms: interventions — Immobilization

STUDY DESIGN:
Intervention Model Description: pragmatic, multi-center, multi-surgeon, prospective outcome study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early pain dependent weight-bearing without immobilization (Experimental): Patients are advised to conduct pain-dependent full weight-bearing starting at the day of study inclusion. In case of severe swelling, a splint or below knee cast can be applied until the initial swelling subsides, but no longer than 14 days. Otherwise, no immobilization is applied. The use of crutches is allowed per the individual patients demands. The physiotherapists at the individual study centers are informed prior to study initiation and are briefed about each patient enrolled in the study. Each patient is handed an information sheet for their outpatient physiotherapist.
  Interventions: Procedure: Early pain dependent weight-bearing without immobilization

INTERVENTIONS:
Procedure: Early pain dependent weight-bearing without immobilization — Patients are advised to conduct pain-dependent full weight-bearing starting at the day of study inclusion. In case of severe swelling, a splint or below knee cast can be applied until the initial swelling subsides, but no longer than 14 days. Otherwise, no immobilization is applied. The use of crutches is allowed per the individual patients demands. The physiotherapists at the individual study centers are informed prior to study initiation and are briefed about each patient enrolled in the study. Each patient is handed an information sheet for their outpatient physiotherapist.

SUMMARY:
The aim of this study is to investigate complication rates and clinical outcome following mobilization and pain-dependent full weight-bearing in a large cohort of patients with surgically treated ankle fractures.

The study design is a pragmatic, multi-center, multi-surgeon, prospective outcome study. Included will be adult patients with any isolated ankle fracture which was treated surgically without additional syndesmotic stabilization (suture-button or syndesmotic screw). Patients included are advised to conduct pain-dependent full weight-bearing without immobilization starting at the day of study inclusion. Follow-up points are 6 weeks, 3-, 6-, and 12 months. Data assessment include radiographic follow-up, complication assessment, return to work/sports, rang of ankle motion, and patient-rated outcome scores (MoxFQ, EFAS, OMAS, EQ-5D-5L). The primary outcomes are complications at 3 months and patient-rated outcome at 12 months. The sample size calculation revealed a final total sample size of 360 patients.

DETAILED DESCRIPTION:
Background Ankle fractures are among the most common fractures in adulthood. Various novel surgical treatment strategies have been developed but nothing has changed regarding the postoperative treatment protocol. Although previous studies indicated that early pain dependent weight-bearing without immobilization in surgically treated ankle fractures is safe, these studies were underpowered.

Therefore, the aim of this pragmatic, multi-center, multi-surgeon, prospective outcome study is to investigate complication rates and clinical outcome following mobilization and pain-dependent full weight-bearing in a large cohort of patients with surgically treated ankle fractures.

Methods The herein proposed study is a pragmatic, multi-center, multi-surgeon, prospective outcome study. Included patients must be independently living and mobile and at least 18 years. Included will be any isolated ankle fracture which was treated surgically without additional syndesmotic stabilization (suture-button or syndesmotic screw). Patients will be recruited following surgical treatment and are advised to conduct pain-dependent full weight-bearing without immobilization starting at the day of study inclusion. The use of crutches is allowed per the individual patients demands. Patients will be invited for follow-up visits at 6 weeks, 3-, 6-, and 12 months. Data assessment at each study point includes radiographic follow-up, complication assessment, return to work/sports, rang of ankle motion, and patient-rated outcome scores (MoxFQ, EFAS, OMAS, EQ-5D-5L). Two primary outcome parameters will be assessed: (1) Complications at 3 months; (2) Patient-rated outcome at 12 months. The sample size calculation revealed a final total sample size of 360 patients. The principle statistical evaluation will be descriptive. For the secondary outcome parameters, a multi-variant regression model will be calculated, individually for complication rates and the patient-rated outcome measures.

Discussion Early pain dependent weightbearing bears the chances to increase patient satisfaction, decrease the time of recovery, and improve the overall patient-rated outcome. These chances must we weighted against a possibly increased risk for complications. Still, the limited data available point at a superiority of early pain-dependent weight-bearing. Due to the high patient number, the herein proposed study is the first to provide resilient data capable of changing the current postoperative rehabilitation regime for surgically treated ankle fractures.

ELIGIBILITY:
Inclusion Criteria:

Patients aged above 18 years Independently living and mobile

Preoperative imaging:

* Unimalleolar fracture: Radiographs in two planes or unilateral CT
* Bi-/Trimalleolar fracture: Unilateral CT Isolated ankle fracture (uni-/ bi-/ trimalleolar fracture)

Surgical treatment:

* Posterior malleolus: Undisplaced fracture: Treatment according to the surgeon's preference; Displaced (≥2mm) fragment of sufficient size (approximately ≥10% of the lateral distal tibia): Open reduction and internal fixation using screw(s) and / or plate(s); Displaced (≥2mm), small fragment (approximately <10% of the lateral distal tibia): Treatment according to the surgeon's preference.
* Lateral malleolus: Open reduction and internal fixation by plate ± compression screw(s).
* Medial malleolus: Closed or open reduction and internal fixation by screw(s) and / or plate(s) osteosynthesis.
* Bony avulsions of the AiTFL (Wagstaffe-Fragment / Tubercule des Chaput): Treatment according to the surgeon's preference.
* Lesions to the Deltoid ligament: Treatment according to the surgeon's preference.
* Arthroscopic assisted fracture treatment: Decision up to the individual surgeon

Postoperative imaging:

* Unimalleolar fracture: Radiographs in two planes or unilateral CT
* Bi-/Trimalleolar fracture: Uni- or bilateral CT Capable of reading and completing the study consent

Exclusion Criteria:

* Age under 18 Surgical stabilization of the distal tibio-fibular joint by syndesmotic screw or dynamic stabilization Concomitant injuries, Charcot neuroarthropathy, pre-existing arthritis, deformity

Tibial pilon fractures, Non-operative treatment

Inability to provide consent, or declining participation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Complications at 3 months follow-up | 3 months +/- 14 Days
  Complications, including surgical side infections, secondary dislocation, or thromboembolic events.
Patient-rated outcome at 12 months follow-up | 12 months +/- 30 days
  Olerud and Mollander Ankle Score (0-100 points; 100=best score)

SECONDARY OUTCOMES:
Patient-rated outcome at 12 months follow-up | 12 months follow-up
  MoXFQ (0-100 metric where 100=most severe)
Patient-rated outcome at 12 months follow-up | 12 months follow-up
  EFAS (0-24 points daily activities, 0-16 points sports scale; 0=worst score)
Patient-rated outcome at 12 months follow-up | 12 months follow-up
  EQ-5D-5L
Fracture characteristics | 3- and 12 months follow-up
  Fracture details, including fracture severity (uni-, bi-, Trimalleolar fractures); comminution, dislocation.
Treatment details | 3- and 12 months follow-up
  Type of osteosynthetic material used, ORIF or AORIF, intra-articular pathologies
Demographics | 3- and 12 months follow-up
  Age, Sex, BMI

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian F Baumbach, MD, Principal Investigator — LMU
Locations (1):
- Department of Trauma Surgery, Medical University of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Patient data will be shared if requested with reasonable arguments.